CLINICAL TRIAL: NCT05247866
Title: Efficacy of Dupilumab on Facilitated Food Introduction in Eosinophilic Esophagitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-019416
Record Dates: First submitted 2021-12-21; First posted 2022-02-21 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: All patients receive active therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Group (Experimental): 30 patients will be given dupilumab (dose based on current approved doses or used in current EoE clinical trial, q weekly dosing) and monitored for clinical response after 12 weeks of therapy)
  Dosing:
  >12 years of age > 40 kg 300 SQ weekly 30- 40 kg 300 mg SQ Q2 weeks 15-29.9 kg 200 mg SQ Q2 weeks
  6-11 years of age 5-15 kg 100 mg SQ Q2W 15-30 kg 200 mg SQ Q2W >30-60 kg 300 mg SQ Q2W
  Interventions: Dietary Supplement: Eosinophilic Esophagitis (EoE) food introduction-1st; Dietary Supplement: Eosinophilic Esophagitis (E0E) food introduction-2nd; Dietary Supplement: Eosinophilic Esophagitis (EoE) Food introduction-3rd dose; Drug: Dupilumab

INTERVENTIONS:
Dietary Supplement: Eosinophilic Esophagitis (EoE) food introduction-1st — 1 serving size of food proven to induce histologic and clinical symptoms in EoE
Dietary Supplement: Eosinophilic Esophagitis (E0E) food introduction-2nd — Either 1 serving size of different food (not food in arm 1) to induce histologic and clinical symptoms in EoE or Increase the food in arm 1 to 2 serving size a day
Dietary Supplement: Eosinophilic Esophagitis (EoE) Food introduction-3rd dose — Either 1 serving size of different food (not food in arm 1 or 2) to induce histologic and clinical symptoms in EoE or Increase the food in arm 2 to 2 serving size a day or unlimited amounts of food arm 1
Drug: Dupilumab — All patients will receive open label dupilumab at the following doses >12 years of age > 40 kg 300 subcutaneous (SQ) weekly
  6-11 years of age 5-15 kg 100 mg SQ every 2 weeks (Q2W) 15-30 kg 200 mg SQ Q2W >30-60 kg 300 mg SQ Q2W

SUMMARY:
Eosinophilic Esophagitis (EoE) is a food driven non-immunoglobulin E (IgE) mediated disease involving eosinophils and type 2 inflammation. Current therapies include diet and the off label use of medications including proton pump inhibitors, topical steroids or biologics. Food elimination creates a decrease quality of life in many children. The goal of the study is to examine a T2 inhibitor (dupilumab) can allow successful reintroduction of allergic EoE foods into the diet. This is a single site study, enrolling subjects 6 to 25 years of age.

DETAILED DESCRIPTION:
This study is an open label exploratory study to examine if patients controlled with dupilumab can successful introduce EoE trigger foods back into their diet.

This is a single site study, enrolling subjects 6 to 25 years of age. In the initial 12 week period, patients will be start on dupilumab on the doses used in the phase 3 trials to control disease. If disease is controlled based on histologic and symptom control at week 12 endoscopy, patients will be start on EoE trigger food. The trigger foods will be based on both a combination of history and histology results. The food will have trigger EoE by histology in the last 2 years and symptoms in the last year when reintroduced into the diet. The study will focus on the the four most common foods that trigger EoE: milk, egg, wheat and soy. For the initial food introduction, the subjects will add one serving size of the food daily for 12 weeks. After 12 weeks, the subjects will have a 2nd endoscopy if the 2nd endoscopy is normal, the subjects will increase the trigger food to 2 serving sizes a day or add an additional trigger food. A 3rd endoscopy will be done if the patients increases the food amount or adds a new food at week 36 (12 weeks after adding the new food). If the subject does not increase or add new foods at week 24, the 3rd endoscopy will not be obtained. All subjects will have end of study endoscopy at week 48.

If the subjects have abnormal endoscopy or increase in symptoms, the amount food will be reduced by 50% and repeat endoscopy will be obtained at the same time schedule-12 weeks later.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 6 to 25 years
2. Diagnosis of Eosinophilic Esophagitis based on the most recent international consensus definition (Dellon et al, Gastroenterology 2019)

   a) History of endoscopy with a peak count of >15 eosinophils per high powered field meeting consensus criteria for Eosinophilic Esophagitis1
3. History of either milk, egg, soy or wheat induced EoE based on the following criteria in the last two years

   1. Addition of a single food lead to exacerbation of esophageal eosinophilia (increase of greater than 15 eos/hpf) or
   2. Removal of a single food lead to normalization of biopsy (esophageal eosinophilia showed less than 6 eos/hpf) AND
   3. History of either milk, egg, soy or wheat induced EoE based on introduction of the food and symptoms in the last 12 months
4. Weight > 10 kg
5. Ability to remain on stable dose of Proton Pump Inhibitor (PPI) therapy throughout the study
6. Girls > 11 years of age must have a negative urine/serum pregnancy test.
7. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Tracheo-esophageal fistulas, inflammatory bowel disease, Barrett's disease, or other significant inflammatory disease of the gastrointestinal tract
2. Biopsy evidence of eosinophilic infiltration in any other organ system
3. History of significant esophageal procedures e.g. sclerotherapy or esophagectomy
4. Systemic immunosuppressant usage in prior 3 months
5. Narrow caliber esophagus defined as the inability to pass a 9.5 mm endoscopy into the esophagus
6. IgE mediated reaction to food (milk, egg, soy or wheat) being introduced in the last 12 months
7. Therapy with biologic molecule (e.g. omalizumab, infliximab) in prior 12 months
8. Any factors that may pose a significant risk for undergoing anesthesia/sedation
9. Subjects undergoing any type of immunotherapy to any food (oral immunotherapy, sublingual immunotherapy, specific oral tolerance induction) within 3 months prior to Visit 1.
10. Active IgE- mediated milk, egg, wheat or soy allergy based on skin test or history (if those foods are being introduced back into the diet).
11. Allergy or known hypersensitivity to the dupilumab.
12. Subjects (or parents of subjects) with obvious excessive anxiety and unlikely to cope with the conditions of an upper Endoscopy and biopsy.
13. Past or current disease(s), which in the opinion of the Investigator or the Sponsor, may affect the subject's participation in this study, including but not limited to active autoimmune disorders, immunodeficiency, malignancy, uncontrolled diseases (hypertension, psychiatric (especially anxiety), cardiac), or other disorders (e.g., liver, gastrointestinal, kidney, cardiovascular, pulmonary disease, or blood disorders).
14. Participation in another clinical intervention study in the three months prior to Visit 1.
15. Subjects unable to follow the protocol and the protocol requirements.
16. Subjects on any experimental drugs or treatments.
17. Subjects unable to read/understand English or follow the protocol and the protocol requirements.
18. Subjects unable to read/understand English or follow the protocol and the protocol requirements.
19. Treatment with a live (attenuated) vaccine within 4 weeks before the baseline visit or throughout the trial
20. Major elective surgeries are prohibited during the study
21. Female patients who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
22. Women of children bearing potential (WOCBP) who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 12 weeks after the last dose. This includes female patients who experience menarche during the study duration and who are unwilling to follow the precautions for WOCBP.
23. Chronic or acute infection requiring treatment with systemic antibiotic, antivirals, or antifungal within 2 weeks of baseline visits

    a. Patients maybe rescreened after infection resolves
24. Participants with active or suspected parasitic infection are excluded.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Spergel, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and published, we will share the study protocol and limited deidentified data.
Supporting Information: Study Protocol
Time Frame: The data will be released after the data is published.

REFERENCES:
- [Background] Rothenberg ME, Dellon ES, Collins MH, Hirano I, Chehade M, Bredenoord AJ, Lucendo AJ, Spergel JM, Sun X, Hamilton JD, Mortensen E, Laws E, Maloney J, Mannent LP, McCann E, Liu X, Glotfelty L, Shabbir A. Efficacy and safety of dupilumab up to 52 weeks in adults and adolescents with eosinophilic oesophagitis (LIBERTY EoE TREET study): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2023 Nov;8(11):990-1004. doi: 10.1016/S2468-1253(23)00204-2. Epub 2023 Aug 31. PMID 37660704
- [Background] McCann E, Chehade M, Spergel JM, Yaworsky A, Symonds T, Stokes J, Tilton ST, Sun X, Kamat S. Validation of the novel Eosinophilic Esophagitis Impact Questionnaire. J Patient Rep Outcomes. 2023 Nov 27;7(1):120. doi: 10.1186/s41687-023-00654-z. PMID 38010430
- [Background] Dellon ES, Rothenberg ME, Collins MH, Hirano I, Chehade M, Bredenoord AJ, Lucendo AJ, Spergel JM, Aceves S, Sun X, Kosloski MP, Kamal MA, Hamilton JD, Beazley B, McCann E, Patel K, Mannent LP, Laws E, Akinlade B, Amin N, Lim WK, Wipperman MF, Ruddy M, Patel N, Weinreich DR, Yancopoulos GD, Shumel B, Maloney J, Giannelou A, Shabbir A. Dupilumab in Adults and Adolescents with Eosinophilic Esophagitis. N Engl J Med. 2022 Dec 22;387(25):2317-2330. doi: 10.1056/NEJMoa2205982. PMID 36546624
- [Background] Spergel BL, Ruffner MA, Godwin BC, Liacouras CA, Cianferoni A, Gober L, Hill DA, Brown-Whitehorn TF, Chaiboonma K, Aceves SA, Muir AM, Spergel JM. Improvement in eosinophilic esophagitis when using dupilumab for other indications or compassionate use. Ann Allergy Asthma Immunol. 2022 May;128(5):589-593. doi: 10.1016/j.anai.2022.01.019. Epub 2022 Jan 25. PMID 35085819
- [Background] Dellon ES, Liacouras CA, Molina-Infante J, Furuta GT, Spergel JM, Zevit N, Spechler SJ, Attwood SE, Straumann A, Aceves SS, Alexander JA, Atkins D, Arva NC, Blanchard C, Bonis PA, Book WM, Capocelli KE, Chehade M, Cheng E, Collins MH, Davis CM, Dias JA, Di Lorenzo C, Dohil R, Dupont C, Falk GW, Ferreira CT, Fox A, Gonsalves NP, Gupta SK, Katzka DA, Kinoshita Y, Menard-Katcher C, Kodroff E, Metz DC, Miehlke S, Muir AB, Mukkada VA, Murch S, Nurko S, Ohtsuka Y, Orel R, Papadopoulou A, Peterson KA, Philpott H, Putnam PE, Richter JE, Rosen R, Rothenberg ME, Schoepfer A, Scott MM, Shah N, Sheikh J, Souza RF, Strobel MJ, Talley NJ, Vaezi MF, Vandenplas Y, Vieira MC, Walker MM, Wechsler JB, Wershil BK, Wen T, Yang GY, Hirano I, Bredenoord AJ. Updated International Consensus Diagnostic Criteria for Eosinophilic Esophagitis: Proceedings of the AGREE Conference. Gastroenterology. 2018 Oct;155(4):1022-1033.e10. doi: 10.1053/j.gastro.2018.07.009. Epub 2018 Sep 6. PMID 30009819
- [Derived] Wolfset N, Muir AB, Benitez AJ, Williams D, De La Torre I, Ruffner MA, Hill DA, Cazeau C, Angello JT, Radwan A, Durrani S, deMarchi S, Spergel JM. Efficacy of Dupilumab on Facilitated Food Reintroduction in Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2025 Sep 30:S1542-3565(25)00745-1. doi: 10.1016/j.cgh.2025.08.025. Online ahead of print. PMID 41038415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 patients recruited
Pre-assignment Details: Open label study, all assigned dupilumab
Period: Overall Study
Arm/Group | Study Group
Started | 21
Completed | 14
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0
Atopy [Number; unit: Count of Participants] — Atopic History
  Count of Participants | 19

OUTCOME MEASURES:

1. Primary Outcome: Esophageal Eosinophilia (Number of Eosinophils in the Esophagus)
Description: Eosinophils per high power field on esophageal biopsy
Time Frame: week 24
Population: 5 patients dropped out to subject withrdraw and anxiety due to injections before completing this endpoint
Measure: Mean (Standard Deviation); unit: eosinophils/high power field
Arm/Group | Study Group
Number analyzed (Participants) | 16
eosinophils/high power field | 5.3 (8.9)

2. Primary Outcome: Esophageal Eosinophilia (Number of Eosinophils in the Esophagus)
Description: Eosinophils per high power field on esophageal biopsy
Time Frame: week 48
Population: 2 patients dropped before this time point
Measure: Mean (Standard Deviation); unit: eosinophils per high power field
Groups:
- Study Group Month 12: 30 patients will be given dupilumab (dose based on current approved doses or used in current EoE clinical trial, q weekly dosing) and monitored for clinical response after 12 weeks of therapy)
  Dosing:
  >12 years of age > 40 kg 300 SQ weekly 30- 40 kg 300 mg SQ Q2 weeks 15-29.9 kg 200 mg SQ Q2 weeks
  6-11 years of age 5-15 kg 100 mg SQ Q2W 15-30 kg 200 mg SQ Q2W >30-60 kg 300 mg SQ Q2W
Arm/Group | Study Group Month 12
Number analyzed (Participants) | 14
eosinophils per high power field | 2.6 (4.5)

3. Primary Outcome: Esophageal Eosinophilia (Number of Eosinophils in the Esophagus)
Description: Eosinophils per high power field on esophageal biopsy
Time Frame: week 36
Measure: Mean (Standard Deviation); unit: eosinophils/high power field
Groups:
- Study Group Month 9: 30 patients will be given dupilumab (dose based on current approved doses or used in current EoE clinical trial, q weekly dosing) and monitored for clinical response after 12 weeks of therapy)
  Dosing:
  >12 years of age > 40 kg 300 SQ weekly 30- 40 kg 300 mg SQ Q2 weeks 15-29.9 kg 200 mg SQ Q2 weeks
  6-11 years of age 5-15 kg 100 mg SQ Q2W 15-30 kg 200 mg SQ Q2W >30-60 kg 300 mg SQ Q2W
Arm/Group | Study Group Month 9
Number analyzed (Participants) | 14
eosinophils/high power field | 1.3 (2.8)

4. Secondary Outcome: Pediatric Eosinophilic Esophagitis Symptom Score (Total Score Based on Pediatric Symptom Score)
Description: Min 0-Max-100, lower is better
Time Frame: week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 16
units on a scale | 7.7 (7.7)

5. Secondary Outcome: Pediatric Eosinophilic Esophagitis Symptom Score (Total Score Based on Pediatric Symptom Score)
Description: Min 0-Max-100, lower is better
Time Frame: week 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 14
units on a scale | 5.1 (6.4)

6. Secondary Outcome: Pediatric Eosinophilic Esophagitis Symptom Score (Total Score Based on Pediatric Symptom Score)
Description: Min 0-Max-100, lower is better
Time Frame: week 48
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 16
units on a scale | 8 (11.3)

7. Other Pre Specified Outcome: Rate of Maintenance of Remission (Less Than <6 Eos/Hpf) in Esophageal Biopsy
Description: Less than 6 eosinophils per high power field in peak count in esophageal biopsy
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 16
Participants | 12

8. Other Pre Specified Outcome: Rate of Maintenance of Remission (Less Than <6 Eos/Hpf) in Esophageal Biopsy
Description: Less than 6 eosinophils per high power field in peak count in esophageal biopsy
Time Frame: week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 14
Participants | 13

9. Other Pre Specified Outcome: Rate of Maintenance of Remission (Less Than <6 Eos/Hpf) in Esophageal Biopsy
Description: Less than 6 eosinophils per high power field in peak count in esophageal biopsy
Time Frame: week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 14
Participants | 11

10. Other Pre Specified Outcome: Rate of Maintenance of Remission (Less Than <15 Eos/Hpf) in Esophageal Biopsy
Description: Less than 15 eosinophils per high power field in peak count in esophageal biopsy
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 16
Participants | 14

11. Other Pre Specified Outcome: Rate of Maintenance of Remission (Less Than <15 Eos/Hpf) in Esophageal Biopsy
Description: Less than 15 eosinophils per high power field in peak count in esophageal biopsy
Time Frame: Week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 14
Participants | 13

12. Other Pre Specified Outcome: Rate of Maintenance of Remission (Less Than <15 Eos/Hpf) in Esophageal Biopsy
Description: Less than15 eosinophils per high power field in peak count in esophageal biopsy
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 14
Participants | 13

13. Other Pre Specified Outcome: Change in Endoscopic Scoring System (EREFS)
Description: Changes from baseline from upper endoscopy validated score (0-10), lower is better
Time Frame: week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 16
units on a scale | 0.6 (0.9)

14. Other Pre Specified Outcome: Change in Endoscopic Scoring System (EREFS)
Description: Changes from baseline from upper endoscopy validated score (0-10), lower is better
Time Frame: week 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 14
units on a scale | 0.4 (0.7)

15. Other Pre Specified Outcome: Change in Endoscopic Scoring System (EREFS)
Description: Changes from baseline from upper endoscopy validated score (0-10), lower is better
Time Frame: week 48
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 14
units on a scale | 0.2 (0.4)

16. Other Pre Specified Outcome: Changes in EoE Quality of Life From Baseline
Description: Changes from baseline in EoE specific Health related Quality of Life (range 0-96), higher is worse
Time Frame: week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 19
units on a scale | 7.06 (6.84)

17. Other Pre Specified Outcome: Changes in EoE Quality of Life From Baseline
Description: Changes from baseline in EoE Health related Quality of Life (range 0-96), higher is worse
Time Frame: week 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 14
units on a scale | 5.14 (6.44)

18. Other Pre Specified Outcome: Changes in EoE Quality of Life From Baseline
Description: Changes from baseline in EoE Health related Quality of Life (range 0-96), higher is worse
Time Frame: week 48
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 14
units on a scale | 8 (11.31)

ADVERSE EVENTS:
Time Frame: Enrollment until end of follow-up (up to 52 weeks)
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=21)
Depression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group (N=21)
headache (Nervous system disorders) | 4
Upper respiratory infection (Infections and infestations) | 8
abdominal Pain (Gastrointestinal disorders) | 4
Injection Reaction (Skin and subcutaneous tissue disorders) | 5
nausea (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 2
Congestion (Respiratory, thoracic and mediastinal disorders) | 2

LIMITATIONS AND CAVEATS:
The study was only completed in pediatrics. If is unclear if the results will extend to adults.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT05247866/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT05247866/ICF_001.pdf